CLINICAL TRIAL: NCT00193401
Title: Phase II Trial of Weekly Topotecan in the First-line Treatment of Elderly Patients With Small Cell Lung Cancer
Brief Title: Weekly Topotecan in the First-line Treatment of Elderly Patients With Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Institutional Review Board TriStar Nashville Market (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 65; 104864665
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Topotecan

INTERVENTIONS:
Drug: Topotecan

SUMMARY:
In this phase II trial, we will evaluate the weekly schedule of topotecan in the first-line treatment of elderly and/or poor performance status patients with extensive stage small cell lung cancer. Patients eligible for this trial will be those considered poor candidates for standard combination chemotherapy or other investigational regimens

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will be receive:

* Topotecan

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Biopsy-proven small cell lung cancer, extensive stage disease
* Age > 65 years
* No previous chemotherapy or radiation therapy.
* Measurable or evaluable disease.
* Adequate bone marrow, liver and kidney function.
* Must be > 4 weeks from previous major surgery
* Must give written informed consent prior to study entry.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Meningeal involvement
* Serious active infections
* Serious underlying medical conditions
* Other active neoplasms

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-08; Primary Completion 2004-06 (Actual); Study Completion 2004-11

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Median survival
1 year and 2 year survival
Overall toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Greco, MD, Principal Investigator — SCRI Development Innovations, LLC